CLINICAL TRIAL: NCT06026254
Title: Rollover Study to Continue IMSA101 Treatments in Patients With Advanced Treatment-Refractory Malignancies Previously Enrolled in the Phase I/IIA Safety and Efficacy Study of IMSA101
Brief Title: A Rollover Study for Subjects Who Completed Participation in IMSA101-101 Trial
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ImmuneSensor Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMSA101-101-R
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination Therapy (Experimental): IMSA101 + ICI
  Interventions: Drug: IMSA101; Drug: Immune Checkpoint Inhibitor

INTERVENTIONS:
Drug: IMSA101 — Intra-tumoral administration on Days 1 and 15 of every 28-day cycle
Drug: Immune Checkpoint Inhibitor — Administered according to product label
  Other Names: ICI

SUMMARY:
This is a rollover study from parent protocol IMSA101-101 for adult patients with advanced malignancies that were previously receiving IMSA101 and who would continue to receive benefit with study treatment of IMSA101 in combination with an immune checkpoint inhibitor (ICI).

DETAILED DESCRIPTION:
The following methodology applies to all patients:

* Treatment cycles will be 28 days in duration with lesions injected every 2 weeks. IMSA101 dose level will remain the same as at the time of the rollover from parent protocol.
* ICI dose level and treatment regimen will remain the same as at the time of the rollover from parent protocol, following the labeled instructions.
* The same single pre-defined lesion/lesion site (longest diameter ≥ 10 mm and ≤ 50 mm) shall be injected throughout study duration, if possible. Where the original injection site is considered by the investigator to become inaccessible, a second lesion/lesion site shall be selected as a replacement and this shall be used henceforth so long as it is considered accessible. Subsequent injection sites shall be replaced when they are considered inaccessible.
* Where no remaining accessible lesions are present and where benefit of IMSA101 therapy is, in the opinion of the investigator, being derived by the patient, continued injections of IMSA101 into the vicinity of an inaccessible lesion or, in the case that a lesion can no longer be radiographically visualized, into the last known location of the non-visible lesion shall be allowed.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and mental capability to understand the informed consent
2. Currently enrolled in parent protocol IMSA101-101 and is receiving IMSA101 treatment
3. Deriving clinical benefit from study treatment, as determined by the investigator
4. Must have fulfilled all required assessments in parent protocol IMSA101-101
5. Male and female patients with reproductive potential must agree to use two forms of highly effective contraception throughout the study

Exclusion Criteria:

1. Permanently discontinued from IMSA101 treatment in parent protocol IMSA101-101 for any reason other than enrollment in the rollover study
2. Failure to meet the criteria specified in parent protocol IMSA101-101 for continued study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Drug-related safety | 12 months
  Frequency of drug-related SAE by subject
Anti-tumor effects | 12 months
  Tumor response based on RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Mooneyham, Study Chair — ImmuneSensor Therapeutics
Locations (2):
- United States (2):
  - Honor Health, Scottsdale, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California

IPD SHARING:
Plan to Share IPD: No